CLINICAL TRIAL: NCT02518971
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of Prophylactic Tamsulosin for Postoperative Urinary Retention in Primary Total Hip and Knee Arthroplasty Patients
Brief Title: Trial of Prophylactic Tamsulosin for Postoperative Urinary Retention in Primary Total Hip and Knee Arthroplasty Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: interim analysis revealed no significant difference between study groups & increased sample size required to gain significance.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Andrew Urquhart, Associate Professor of Orthopaedic Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00087825
Record Dates: First submitted 2015-07-27; First posted 2015-08-10 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Urinary Retention
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- tamsulosin (Experimental): 0.4 mg daily for five days pre-op through post-op day one (seven total)
  Interventions: Drug: Tamsulosin
- placebo (Placebo Comparator): One capsule daily for five days pre-op through post-op day one (seven total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — 0.4 mg daily
  Other Names: Flomax
  Arms: tamsulosin
Drug: Placebo — one capsule daily
  Arms: placebo

SUMMARY:
The study aims to evaluate the efficacy of prophylactic tamsulosin in reducing the incidence of postoperative urinary retention in primary total knee and hip arthroplasty patients.

DETAILED DESCRIPTION:
Prophylactic administration of tamsulosin will be compared to a placebo to evaluate the effectiveness in reducing the incidence of postoperative urinary retention in total hip and knee arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* Men age 35 or older
* Primary total hip and knee arthroplasty patients (general, spinal, or epidural anesthesia
* No current use (>1 month) of alpha-blockers
* Community ambulator
* Adequate organ and marrow function as defined below:

leucocytes at least 3,000/µL, absolute neutrophil count at least 1,500/µL, platelets at least 100,000/µL, creatinine within normal institutional limits

* Ability to understand, and the willingness to sign, a written informed consent

Exclusion Criteria:

* History of radical prostatectomy
* Receiving any other investigational agents
* Revision hip and knee arthroplasty patients
* Severe liver or kidney disease
* Taking strong inhibitors of CYP3A4 (ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir/ritonavir, lopinavir, or conivaptan)
* Being on alpha-blockers (alfuzosin, doxazosin, prazosin, terazosin, tamsulosin, phenoxybenzamine, or silodosin)
* Being of 5-alpha reductase inhibitors (finasteride, dutasteride)
* History of allergy or sensitivity to tamsulosin or other alpha-blockers (alfuzosin, doxazosin, prazosin, terazosin, or phenoxybenzamine)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Taking Sildenafil,Tadalafil, or Vardenafil

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Urquhart, MD, Principal Investigator — University of Michigan, Dept of Orthopaedic Surgery; Manuel Schubert, MD, Study Director — University of Michigan, Dept of Orthopaedic Surgery
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 176 subjects were enrolled in the study. 174 were randomized to either the active tamsulosin group or placebo group and 2 subjects were withdrawn prior to randomization. 43 additional patients were withdrawn after randomization.
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 87 | 87
Completed | 64 | 67
Not Completed | 23 | 20
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 6 | 6
Not completed — Protocol Violation | 6 | 4
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Side effects | 1 | 0
Not completed — medication lost in mail | 0 | 1
Not completed — eligibility criteria no longer met | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 64 | 67 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.55 (10.4) | 61.37 (9.6) | 60.98 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 64 | 67 | 131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients to Develop Postoperative Urinary Retention (POUR)
Description: Patients who have not developed POUR will have two consecutive, spontaneous urine voids with residual volume of less than 200 mL, as determined by bladder scan or straight catheterization. Patients who do not successfully have the two spontaneous urine voids of less than 200 mL will be considered as having developed POUR. The incidence of POUR will be compared statistically between those taking and not taking tamsulosin at the time of surgery.
Time Frame: Postop day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 67
Participants | 18 | 24
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Other; p = 0.345, Chi-squared

2. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay will be recorded in days and compared statistically between the two groups .
Time Frame: 1-4 days postoperative
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 67
days | 1.125 (0.42) | 1.209 (0.64)
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Other; p = .378, Student T-Test

3. Secondary Outcome: Incidence of Discharge to a Skilled Nursing Facility
Description: Discharge to a skilled nursing facility will be recorded (yes/no) and compared statistically between the two groups.
Time Frame: 1-4 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 67
Participants | 1 | 1
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Other; p = 1.0, Fisher Exact

4. Secondary Outcome: Incidence of Surgical Site Infection
Description: Surgical site infection will be recorded (yes/no) and compared statistically between the two groups.
Time Frame: Up to two weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 64
Participants | 0 | 2
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Other; p = .497, Fisher Exact

5. Secondary Outcome: Acute Postoperative Pain Medication Dosages
Description: The dosages of postoperative pain medications will be compared statistically between the two groups.
Time Frame: Postoperative day 1 to day of discharge (1-4 days on average)
Measure: Mean (Standard Deviation); unit: morphine equivalent doses
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 67
morphine equivalent doses | 44.85 (47.18) | 36 (31.56)
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Other; p = .207, Student T-test

6. Secondary Outcome: Incidence of Postoperative Complications
Description: Postoperative complications will be recorded and the incidence will be compared statistically between the two groups.
Time Frame: Up to 31 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 64 | 67
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 31 days post-operatively
Groups:
- Not Randomized: Participants were withdrawn from study before randomization
Arm/Group | Tamsulosin | Placebo | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/67 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/64 | 0/67 | 0/2
Other Adverse Events (participants affected / at risk) | 20/64 | 11/67 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=64) | Placebo (N=67) | Not Randomized (N=2)
Floppy Iris Syndrome (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=64) | Placebo (N=67) | Not Randomized (N=2)
hypotension (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (General disorders) | 1 (1) | 2 (2) | 0 (0)
Syncope (General disorders) | 3 (3) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
increased post operative pain (Surgical and medical procedures) | 5 (5) | 2 (2) | 0 (0)
delayed wound healing/wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical Site Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Calf Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Hives/pruritus (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Altered Mental Status (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gout Flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02518971/Prot_SAP_000.pdf